CLINICAL TRIAL: NCT07202442
Title: Beginning of Robotic Emergency General Surgery Program at Nice University Hospital
Brief Title: Robotic Emergency General Surgery Program
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Urgences01
Record Dates: First submitted 2025-09-19; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Emergency General Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Emergency General surgery patients with robotic approach for the surgery — vPrimary Endpoint: The proportion of procedures performed robotically versus laparoscopically or via laparotomy for selected indications. Secondary Endpoints: A 5% change in perioperative morbidity, laparotomy rate, LOS, critical care admission rate, and operative time. Included Pathologies (for patients eligible for laparoscopy) : Acute cholecystitis with predictors of intraoperative difficulty. Bowel obstruction requiring bowel resection (in presence of CT signs of visceral compromise: poor enhancement of bowel loops, pneumoperitoneum). Complicated acute diverticulitis with perforation and peritonitis. Penetrating abdominal trauma with hemodynamic stability requiring surgery (e.g., bowel resection-anastomosis). Right or left colectomy for other etiologies. Splenectomy in hemodynamically stable or embolized patients.

SUMMARY:
Background Abdominal surgical emergencies account for 20-30% of visceral surgery procedures. However, these emergencies are responsible for more than half of the morbidity in our discipline, with a surgical site infection rate four times higher than in elective surgery, and significantly higher rates of surgical revision and conversion (PMID: 34225343 and 27016997 and 27120712). In cases where minimally invasive surgery is converted to laparotomy, patients are three times more likely to be admitted to critical care units (PMID: 39966134). Visceral surgery currently represents the largest and fastest-growing discipline in robotic surgery. Robotic management of emergency general surgery has been described in the literature for several years, particularly in the United States. Robotic surgery allows a shift from open procedures to minimally invasive techniques or simplifies complex laparoscopic procedures. Several literature reviews and meta-analyses report decreased laparotomy rates, reduced perioperative morbidity, and shorter average length of hospital stay (PMID: 38446451 and 38918109). Abdominal surgical emergencies account for 20-30% of visceral surgery procedures. However, these emergencies are responsible for more than half of the morbidity in our discipline, with a surgical site infection rate four times higher than in elective surgery, and significantly higher rates of surgical revision and conversion (PMID: 34225343 and 27016997 and 27120712). In cases where minimally invasive surgery is converted to laparotomy, patients are three times more likely to be admitted to critical care units (PMID: 39966134). Visceral surgery currently represents the largest and fastest-growing discipline in robotic surgery. Robotic management of emergency general surgery has been described in the literature for several years, particularly in the United States. Robotic surgery allows a shift from open procedures to minimally invasive techniques or simplifies complex laparoscopic procedures. Several literature reviews and meta-analyses report decreased laparotomy rates, reduced perioperative morbidity, and shorter average length of hospital stay (PMID: 38446451 and 38918109).Primary Objective:To assess the implementation of a robotic surgery program for emergency visceral procedures (proof of feasibility in our university hospital). Secondary Objectives: Reduce perioperative morbidity, Reduce the rate of laparotomy, Reduce the average length of hospital stay (LOS), Reduce postoperative admission to critical care, Reduce operative time.

ELIGIBILITY:
Inclusion Criteria:

* Acute cholecystitis with predictors of intraoperative difficulty.
* Bowel obstruction requiring bowel resection (in presence of CT signs of visceral compromise: poor enhancement of bowel loops, pneumoperitoneum).
* Complicated acute diverticulitis with perforation and peritonitis.
* Penetrating abdominal trauma with hemodynamic stability requiring surgery (e.g., bowel resection-anastomosis).
* Right or left colectomy for other etiologies.
* Splenectomy in hemodynamically stable or embolized patients.

Exclusion Criteria:

* Hemodynamic instability.
* Uncomplicated acute appendicitis.
* Acute cholecystitis without predictors of intraoperative difficulty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency general surgery patients admitted to Nice University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Implementation of a robotic surgery program for emergency visceral procedures | Postoperative day 30
  To assess the implementation of a robotic surgery program for emergency visceral procedures (proof of feasibility in our university hospital).The team will screen patients who will meet the inclusion criteria and the first score will be : were we able to purpose robotic approach fr the patient. Then if we were able to do it, and if not, the reason why (OT nurse difficulty ? technical issue ? other ?).

SECONDARY OUTCOMES:
Evaluating robotic general emergencies procedures (Change perioperative morbidity) | Postoperative day 30.
  Clavien-Dindo Classification ( grade 1 to 5) vs an historical cohort
Evaluating robotic general emergencies procedures (Change the rate of laparotomy) | Postoperative day 30
  Pourcentage vs historical data
Evaluating robotic general emergencies procedures (Change the average length of hospital stay ) | Postoperative day 30
  (LOS)-(in days, vs historical data)
Evaluating robotic general emergencies procedures (Change postoperative admission to critical care) | Postoperative day 30
  Pourcentage vs historical data
Evaluating robotic general emergencies procedures (Change operative time) | Postoperative day 30
  In minutes, vs historical data

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, Alpes Maritimes, France